CLINICAL TRIAL: NCT07016087
Title: Therapeutic Efficacy of Cutaneous Application of Postbiotic N-(1-carbamoyl-2-phenyl-ethyl) Butyramide (FBA) in Pediatric Subjects Affected by Atopic Dermatitis - BuPAD Trial (Butyrate for Pediatric Atopic Dermatitis)
Brief Title: Therapeutic Efficacy of Cutaneous Application of Postbiotic N-(1-carbamoyl-2-phenyl-ethyl) Butyramide (FBA) in Pediatric Subjects Affected by Atopic Dermatitis
Acronym: BuPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, MD,PhD,Prof, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 102/24
Record Dates: First submitted 2025-05-21; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): AD affected patients treated with butyrate-free emollients
  Interventions: Other: Cosmetic formulation usual
- Group B (Experimental): AD affected patients treated with emollients added with butyrate releaser
  Interventions: Other: Cosmetic formulation experimental

INTERVENTIONS:
Other: Cosmetic formulation experimental — Cosmetic formulation containing emollients and a butyrate releaser: the postbiotic N-(1-carbamoyl-2-phenyl-ethyl) butyramide (FBA)
  Arms: Group B
Other: Cosmetic formulation usual — Cosmetic formulation containing emollients
  Arms: Group A

SUMMARY:
Atopic dermatitis (AD) is a chronic, multifactorial inflammatory skin disease characterized by eczematous skin and pruritus and it's due to an alteration of the skin barrier and of the intestinal and skin microbiome (SM), which normally contributes to maintaining skin integrity and modulating host inflammatory responses. This alteration leads to a lower production of butyrate, a short-chain fatty acid capable of reducing skin permeability by improving barrier integrity, performing a trophic effect on the skin and suppressing local inflammatory responses. Furthermore, a reduction of butyrate in patients with AD has also been demonstrated at the intestinal level.

Conventional therapy for AD consists of eliminating exacerbating factors, applying emollients and in exacerbations, or in moderate/severe forms, applying topical steroids or topical calcineurin inhibitors. The possibility of using emollients containing substances physiologically present in the skin, such as butyrate, could represent a safe treatment strategy, capable of reducing exacerbations and therefore the evolution towards moderate-severe forms of AD.

On the basis of these premises, the BuPad study aims to evaluate the therapeutic efficacy of the cutaneous application of a butyrate releaser, the postbiotic N-(1-carbamoyl-2-phenyl-ethyl) butyramide (FBA) in a cosmetic formulation, in children affected by AD.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Age: 6-36 months
* Caucasian ethnicity
* Diagnosis of atopic dermatitis
* Written informed consent of parents/legal guardians

Exclusion Criteria:

* Age <6 months and >36 months
* non-Caucasian ethnicity
* skin infections
* ichthyosis
* food allergies
* chronic systemic diseases
* congenital heart defects
* tuberculosis
* autoimmune disorders
* immunodeficiency
* inflammatory bowel disease
* celiac disease
* cystic fibrosis
* metabolic disorders
* neoplasms
* chronic pulmonary disorders
* gastrointestinal tract malformations
* respiratory tract malformations
* intake of systemic prebiotics/probiotics/synbiotics/immunomodulators 4 weeks prior to enrollment
* treatment with topical immunomodulators (Tacrolimus or Pimecrolimus) within 3 months prior to enrollment
* use of topical or systemic corticosteroids or calcineurin antagonists or phototherapy within the previous 4 weeks
* investigator uncertainty about the subject's willingness or ability to comply with protocol requirements
* participation in any other study involving investigational or marketed products concurrently or within two weeks prior to study entry hypersensitivity to any component of the investigational product
* absence of written informed consent

Ages: 6 Months to 26 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of topical therapy with a butyrate releaser in children with AD | At 12 weeks
  Evaluation of the efficacy of topical therapy with a butyrate releaser in children with AD by reduction of SCORAD index after 12 weeks of treatment (T12).

SECONDARY OUTCOMES:
Changes in the SCORAD index | At baseline, at 4 weeks, at 8 weeks, at 12 weeks, at 16 weeks
  Mean changes in the SCORAD index comparing the baseline value (T0) and the values after 4 weeks (T4) and 8 weeks (T8) of treatment and 4 weeks after the end of treatment (T16)
Changes in Transepidermal Water Loss (TEWL) | At baseline, at 4 weeks, at 8 weeks, at 12 weeks, at 16 weeks
  Mean changes in Transepidermal Water Loss (TEWL) comparing the baseline value (T0) and the values after 4 weeks (T4), 8 weeks (T8) and 12 weeks of treatment (T12) and 4 weeks after the end of treatment (T16)
Assessment of skin microbiota | At baseline, at 12 weeks
  Assessment of the skin microbiota composition at baseline (T0) and at the end of treatment (T12)
Number of skin infections during the study period | At 16 weeks
  Number of skin infections during the study period (last follow up after 16 weeks from the start of treatment)
Days without use of cortisone | At 12 weeks, at 16 weeks
  Assessment of days without use of cortisone at T12 and at T16
Infant Dermatitis Quality of Life Questionnaire (IDQOL) | At baseline, at 4 weeks, at 8 weeks, at 12 weeks, at 16 weeks
  Mean changes in the Infant Dermatitis Quality of Life Questionnaire (IDQOL) at T0, T4, T8, T12, T16

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy